CLINICAL TRIAL: NCT03834493
Title: A Phase 3, Randomized, Double-blind Trial of Pembrolizumab (MK-3475) Plus Enzalutamide Versus Placebo Plus Enzalutamide in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC) (KEYNOTE-641)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Enzalutamide Versus Placebo Plus Enzalutamide in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-3475-641/KEYNOTE-641)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-641; MK-3475-641 (Other: Merck Protocol Number); KEYNOTE-641 (Other: Merck); 195005 (Registry Identifier: JAPIC-CTI); 2022-500785-10-00 (Registry Identifier: EU CT); U1111-1278-1151 (Registry Identifier: UTN); 2018-004117-40 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Prostatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enzalutamide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study became unblinded in February 2023.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Enzalutamide (Experimental): Participants receive 200 mg pembrolizumab by intravenous (IV) infusion administered on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 2 years) PLUS enzalutamide 160 mg administered orally (PO) once a day (QD) continuously until progression.
  Interventions: Biological: Pembrolizumab; Drug: Enzalutamide
- Placebo + Enzalutamide (Placebo Comparator): Participants receive placebo by IV infusion administered on Day 1 Q3W for up to 35 cycles (approximately 2 years) PLUS enzalutamide 160 mg administered PO QD continuously until progression.
  Interventions: Drug: Enzalutamide; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + Enzalutamide
Drug: Enzalutamide — Capsules/Tablets
  Other Names: XTANDI®
Drug: Placebo — IV infusion
  Other Names: Normal saline or dextrose infusion
  Arms: Placebo + Enzalutamide

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of pembrolizumab (MK-3475) and enzalutamide in the treatment of men with metastatic castration-resistant prostate cancer (mCRPC) who have not received chemotherapy for mCRPC, are abiraterone-naïve, or are intolerant to or progressed on abiraterone acetate. There are two primary study hypotheses.

Hypothesis 1: The combination of pembrolizumab plus enzalutamide is superior to placebo plus enzalutamide with respect to Overall Survival (OS).

Hypothesis 2: The combination of pembrolizumab plus enzalutamide is superior to placebo plus enzalutamide with respect to Radiographic Progression-free Survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while on androgen deprivation therapy (or post bilateral orchiectomy) within 6 months prior to randomization
* Has current evidence of metastatic disease documented by either bone lesions on bone scan and/or soft tissue disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Has met one of the following criteria with regard to abiraterone acetate exposure: (1) is abiraterone-naïve; (2) received prior abiraterone acetate for the treatment of mHSPC or mCRPC, for a minimum of 4 weeks and not progressed while on treatment; or (3) received prior abiraterone acetate for the treatment of mHSPC or mCRPC and progressed on treatment after a minimum of 8 weeks treatment (minimum 14 weeks for those with bone progression)
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM)
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses prior to randomization
* Participants must agree to the following during the study treatment period and for at least 90 days after the last dose of enzalutamide: Refrain from donating sperm, plus EITHER be abstinent OR must agree to use male condom
* Has provided newly obtained core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed). Participants with bone only or bone predominant disease may provide a bone biopsy sample
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to randomization and not recovered adequately from the toxicities and/or complications
* Has a gastrointestinal disorder affecting absorption or is unable to swallow tablets/capsules
* Has an active infection (including tuberculosis) requiring systemic therapy
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease
* Has known active human immunodeficiency virus (HIV), concurrent active hepatitis B virus (HBV) or known active hepatitis C virus (HCV) infection
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has hypersensitivity to pembrolizumab and/or enzalutamide and/or any of their excipients
* Has a history of seizure or any condition that may predispose to seizure
* Has a history of loss of consciousness within 12 months of screening
* Has hypotension (systolic blood pressure <86 millimeters of mercury [mmHg]) or uncontrolled hypertension (systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg) at the screening visit
* Has bradycardia (heart rate of <50 beats per minute) on the screening electrocardiogram (ECG)
* Has history of prostate cancer progression on ketoconazole
* Has had prior treatment with enzalutamide, apalutamide, darolutamide or cytochrome P450 (CYP) 17 inhibitor other than abiraterone acetate
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received prior treatment with radium or other therapeutic radiopharmaceuticals for prostate cancer
* Has received prior treatment with docetaxel or another chemotherapy agent for mCRPC
* Has had a prior anti-cancer monoclonal antibody (mAb) prior to randomization
* Has used herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (eg, saw palmetto) prior to randomization
* Has received a live or live attenuated vaccine within 30 days prior to randomization
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a "superscan" bone scan
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 90 days after the last dose of enzalutamide
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1244 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2026-05-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (259):
- United States (28):
  - University of South Alabama, Mitchell Cancer Institute ( Site 0065), Mobile, Alabama
  - Providence Medical Foundation-Oncology ( Site 0069), Fullerton, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0081), Los Angeles, California
  - University of Colorado Cancer Center ( Site 0022), Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven ( Site 0038), New Haven, Connecticut
  - Moffitt Cancer Center ( Site 0080), Tampa, Florida
  - Georgia Cancer Center at Augusta University ( Site 0026), Augusta, Georgia
  - Mount Sinai Hospital ( Site 0042), Chicago, Illinois
  - Methodist Hospitals. ( Site 0008), Merrillville, Indiana
  - Tulane Cancer Center ( Site 0066), New Orleans, Louisiana
  - University of Massachusetts Worcester ( Site 0053), Worcester, Massachusetts
  - Cancer & Hematology Centers of Western Michigan ( Site 0013), Grand Rapids, Michigan
  - Munson Medical Center ( Site 0030), Traverse City, Michigan
  - St. Vincent Frontier Cancer Center ( Site 0016), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 0034), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada ( Site 0092), Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0004), Hackensack, New Jersey
  - Associated Medical Professionals of NY ( Site 0060), Syracuse, New York
  - W. G. Bill Hefner VA Medical Center ( Site 0029), Salisbury, North Carolina
  - Gabrail Cancer Center-Research ( Site 0096), Canton, Ohio
  - Tri-State Urologic Services PSC, Inc. ( Site 0094), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 0036), Cleveland, Ohio
  - Oregon Health Science University ( Site 0031), Portland, Oregon
  - Carolina Urologic Research Center ( Site 0070), Myrtle Beach, South Carolina
  - Inova Schar Cancer Institute ( Site 0006), Fairfax, Virginia
  - Virginia Cancer Institute ( Site 0052), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0086), Roanoke, Virginia
  - Froedtert Hospital & the Medical College of Wisconsin ( Site 0045), Milwaukee, Wisconsin
- Argentina (13):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 1013), Berazategui, Buenos Aires
  - Organizacion Medica de Investigacion ( Site 1019), CABA, Buenos Aires
  - Instituto Medico Alexander Fleming ( Site 1010), Ciudad Autonoma de Buenos Aires., Buenos Aires
  - Instituto de Investigaciones Clinicas ( Site 1000), Mar del Plata, Buenos Aires
  - Centro de Diagnostico Urologico ( Site 1008), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 1002), Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario ( Site 1015), Rosario, Santa Fe Province
  - Instituto de Investigaciones Metabolicas [Buenos Aires, Argentina] ( Site 1011), Buenos Aires
  - Hospital Aleman ( Site 1004), Buenos Aires
  - Centro Medico Dra De Salvo ( Site 1018), Buenos Aires
  - CEMAIC ( Site 1014), Córdoba
  - Centro Oncologico Riojano Integral ( Site 1005), La Rioja
  - Centro Oncologico de Integracion Regional. COIR ( Site 1007), Mendoza
- Australia (10):
  - St. Vincent's Hospital ( Site 0158), Darlinghurst, New South Wales
  - St George Hospital ( Site 0157), Kogarah, New South Wales
  - Macquarie University ( Site 0151), Macquarie University, New South Wales
  - Port Macquarie Base Hospital ( Site 0153), Port Macquarie, New South Wales
  - Calvary Mater Newcastle ( Site 0148), Waratah, New South Wales
  - Gallipoli Medical Research Ltd ( Site 0149), Greenslopes, Queensland
  - Gold Coast University Hospital ( Site 0150), Southport, Queensland
  - Royal Adelaide Hospital ( Site 0154), Adelaide, South Australia
  - Monash Medical Centre ( Site 0147), Clayton, Victoria
  - Fiona Stanley Hospital ( Site 0162), Perth, Western Australia
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 0373), Linz, Upper Austria
  - Medizinische Universität Wien ( Site 0375), Vienna
- Brazil (8):
  - Hospital Erasto Gaertner-CEPEP - Pesquisa Clínica ( Site 1036), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 1032), Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 1038), Ijuí, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 1021), Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 1035), Itajaí, Santa Catarina
  - Hospital de Base de Sao Jose de Rio Preto ( Site 1022), São José do Rio Preto, São Paulo
  - A.C. Camargo Cancer Center ( Site 1026), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 1040), São Paulo
- Bulgaria (3):
  - MHAT Serdika-Second Department of Medical Oncology ( Site 0505), Sofia, Sofia (stolitsa)
  - MHAT Central Hospital ( Site 0503), Plovdiv
  - Complex Cancer Center Plovdiv-First Medical Oncology Department ( Site 0507), Plovdiv
- Canada (12):
  - BC Cancer Victoria-Clinical Trials Unit ( Site 0111), Victoria, British Columbia
  - Health Sciences North ( Site 0122), Greater Sudbury, Ontario
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0116), Hamilton, Ontario
  - Grand River Hospital ( Site 0120), Kitchener, Ontario
  - Lakeridge Health ( Site 0117), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 0108), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0107), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0119), Greenfield Park, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0106), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0103), Québec, Quebec
  - CIUSSS du Bas Saint Laurent - Hopital Regional de Rimouski ( Site 0102), Rimouski, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0105), Sherbrooke, Quebec
- Chile (6):
  - Fundacion Arturo Lopez Perez ( Site 1049), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1047), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 1044), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1041), Temuco, Región de la Araucanía
  - Rey y Oreilly Limitada ( Site 1048), Temuco, Región de la Araucanía
  - Oncocentro ( Site 1045), Viña del Mar, Región de Valparaíso
- Colombia (8):
  - Hospital Pablo Tobon Uribe ( Site 1066), Medellín, Antioquia
  - Biomelab S A S ( Site 1067), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 1073), Barranquilla, Atlántico
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 1062), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 1068), Valledupar, Cesar Department
  - Oncomédica S.A.S ( Site 1057), Montería, Departamento de Córdoba
  - Clínica Imbanaco S.A.S ( Site 1064), Cali, Valle del Cauca Department
  - Hemato Oncologos S.A. ( Site 1065), Cali, Valle del Cauca Department
- Czechia (3):
  - Fakultni Nemocnice u sv. Anny v Brne-Onkologicko-chirurgicke oddeleni ( Site 1303), Brno, Brno-mesto
  - Nemocnice AGEL Novy Jicin a.s. ( Site 1304), Nový Jičín, Novy Jicin
  - Fakultni nemocnice Olomouc ( Site 1301), Olomouc, Olomoucký kraj
- France (18):
  - C.H. de Saint Quentin ( Site 0481), Saint-Quentin, Aisne
  - Centre Jean Perrin ( Site 0434), Clermont-Ferrand, Auvergne
  - Clinique Sainte Anne ( Site 0431), Strasbourg, Bas-Rhin
  - CHU de Brest -Site Hopital Morvan ( Site 0441), Brest, Brittany Region
  - CHU Jean Minjoz ( Site 0423), Besançon, Doubs
  - Institut Bergonie ( Site 0421), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0418), Toulouse, Haute-Garonne
  - Hopital Foch ( Site 0428), Suresnes, Hauts-de-Seine
  - Institut Regional du Cancer de Montpellier - ICM ( Site 0443), Montpellier, Herault
  - Institut De Cancerologie De L Ouest ( Site 0448), Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Regional du Orleans ( Site 0430), Orléans, Loiret
  - Centre D Oncologie de Gentilly ( Site 0432), Nancy, Meurthe-et-Moselle
  - Centre Hospitalier de Valenciennes ( Site 0439), Valenciennes, Nord
  - C.H.U. Lyon Sud ( Site 0436), Pierre-Bénite, Rhone
  - CHU Amiens Picardie Site Sud Amiens ( Site 0438), Amiens, Somme
  - Institut Gustave Roussy ( Site 0416), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 0447), Avignon, Vaucluse
  - Institut Mutualiste Montsouris ( Site 0446), Paris
- Germany (13):
  - Universitaetsklinikum Freiburg - Medizinische Klinik ( Site 0304), Freiburg im Breisgau, Baden-Wurttemberg
  - Studienpraxis Urologie ( Site 0309), Nürtingen, Baden-Wurttemberg
  - Universitaetsklinik fuer Urologie ( Site 0307), Tübingen, Baden-Wurttemberg
  - Klinikum Rechts der Isar ( Site 0300), Munich, Bavaria
  - Universitaetsklinik der Paracelsus Medizinischen Privatuniversitaet ( Site 0318), Nuremberg, Bavaria
  - Universitaetsklinikum Goettingen ( Site 0345), Göttingen, Lower Saxony
  - Uniklinik RWTH Aachen ( Site 0308), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0320), Münster, North Rhine-Westphalia
  - Krankenhaus der Barmherzigen Brueder Trier ( Site 0310), Trier, Rhineland-Palatinate
  - Universitaetsklinikum des Saarlandes ( Site 0348), Homburg, Saarland
  - Universitaetsklinikum Schleswig Holstein. ( Site 0346), Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Jena ( Site 0305), Jena, Thuringia
  - Charite Universitaetsmedizin Berlin ( Site 0301), Berlin
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1321), Kecskemét, Bács-Kiskun county
  - Petz Aladár Megyei Oktató Kórház-Onkológiai Osztály ( Site 1324), Győr, Győr-Moson-Sopron
  - Országos Onkológiai Intézet-Urogenital Tumors Department and Clinical Pharmacology ( Site 1325), Budapest, Pest County
  - Magyar Honvedseg Egeszsegugyi Kozpont-Onkologiai Osztaly ( Site 1326), Budapest
- Ireland (3):
  - Beaumont Hospital ( Site 0726), Dublin
  - Tallaght University Hospital ( Site 0730), Dublin
  - Mid Western Cancer Centre ( Site 0728), Limerick
- Israel (10):
  - HaEmek Medical Center ( Site 0548), Afula
  - Assuta Ashdod Medical Center ( Site 0550), Ashdod
  - Soroka Medical Center ( Site 0549), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0543), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0546), Jerusalem
  - Meir Medical Center ( Site 0544), Kfar Saba
  - Rabin Medical Center ( Site 0545), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0541), Ramat Gan
  - Sourasky Medical Center ( Site 0542), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0547), Ẕerifin
- Italy (14):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-Oncologia Medica ( Site 0464), Meldola, Emilia-Romagna
  - A.O. Universitaria di Modena ( Site 0454), Modena, Emilia-Romagna
  - Istituto Clinico Humanitas Research Hospital ( Site 0452), Rozzano, Lombardy
  - Presidio Ospedaliero S. Maria Delle Grazie-U.O.C. ONCOLOGIA ( Site 0802), Pozzuoli, Napoli
  - Centro Di Riferimento Oncologico ( Site 0800), Aviano, Pordenone
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma-Oncology Unit ( Site 0465), Verona, Veneto
  - Medical Oncology Ospedale San Donato ( Site 0461), Arezzo
  - Ospedale Policlinico S. Orsola-Malpighi ( Site 0453), Bologna
  - Azienda Ospedaliera Cannizzaro ( Site 0458), Catania
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0462), Napoli
  - Azienda Ospedaliera San Camillo Forlanini ( Site 0455), Roma
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 0801), Roma
  - Azienda Ospedaliera Santa Maria Terni ( Site 0456), Terni
  - Az. Osp. Univ. Sta Maria della Misericordia di Udine ( Site 0460), Udine
- Japan (25):
  - National Cancer Center Hospital East ( Site 0702), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 0703), Sakura, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0716), Matsuyama, Ehime
  - Iizuka Hospital ( Site 0744), Iizuka, Fukuoka
  - Hakodate Goryoukaku Hospital ( Site 0739), Hakodate, Hokkaido
  - Kanazawa University Hospital ( Site 0701), Kanazawa, Ishikawa-ken
  - Kitasato University Hospital ( Site 0705), Sagamihara, Kanagawa
  - Yokohama City University Medical Center ( Site 0706), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 0747), Natori-shi, Miyagi
  - Nara Medical University Hospital ( Site 0715), Kashihara, Nara
  - Kindai University Hospital ( Site 0714), Sayama, Osaka
  - The University of Osaka Hospital ( Site 0713), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 0708), Hidaka, Saitama
  - Saitama Medical Center ( Site 0743), Kawagoe, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 0707), Koshigaya, Saitama
  - Hamamatsu University Hospital ( Site 0720), Hamamatsu, Shizuoka
  - Yamaguchi University Hospital ( Site 0717), Ube, Yamaguchi
  - Chiba Cancer Center ( Site 0704), Chiba
  - Kyushu University Hospital ( Site 0718), Fukuoka
  - Hiroshima Prefectural Hospital ( Site 0748), Hiroshima
  - University of Miyazaki Hospital ( Site 0721), Miyazaki
  - Nagasaki University Hospital ( Site 0719), Nagasaki
  - Toranomon Hospital ( Site 0711), Tokyo
  - Nippon Medical School Hospital ( Site 0709), Tokyo
  - Keio University Hospital ( Site 0710), Tokyo
- Netherlands (11):
  - Radboud University Medical Center ( Site 0470), Nijmegen, Gelderland
  - Maastricht University Medical Centre ( Site 0467), Maastricht, Limburg
  - Amphia Hospital Location Molengracht ( Site 0474), Breda, North Brabant
  - Catharina Ziekenhuis ( Site 0472), Eindhoven, North Brabant
  - Noordwest Ziekenhuisgroep NWZ ( Site 0468), Alkmaar, North Holland
  - Vrije Universiteit Medisch Centrum ( Site 0479), Amsterdam, North Holland
  - Tergooiziekenhuizen ( Site 0466), Hilversum, North Holland
  - Spaarne Ziekenhuis ( Site 0473), Hoofddorp, North Holland
  - Ziekenhuisgroep Twente ( Site 0469), Hengelo, Overijssel
  - Haaglanden MC - locatie Antoniushove ( Site 0471), Leidschendam, South Holland
  - Franciscus Gasthuis en Vlietland ( Site 0489), Schiedam, South Holland
- New Zealand (3):
  - Tauranga Hospital ( Site 0215), Tauranga, Bay of Plenty
  - Canterbury Regional Cancer & Blood Service ( Site 0195), Christchurch, Canterbury
  - Auckland City Hospital ( Site 0193), Auckland
- Poland (6):
  - Przychodnia Lekarska Komed ( Site 0628), Konin, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 0636), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Clinical Best Solutions ( Site 0622), Warsaw, Masovian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 0624), Koszalin, West Pomeranian Voivodeship
  - Salve Medica SP ( Site 0686), Lodz, Łódź Voivodeship
  - Provita Prolife Centrum Medyczne ( Site 0630), Tomaszów Mazowiecki, Łódź Voivodeship
- Puerto Rico (2):
  - Puerto Rico Medical Research Center LLC ( Site 1122), San Juan
  - FDI Clinical Research ( Site 1121), San Juan
- Russia (10):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 0565), Chelyabinsk, Chelyabinsk Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0585), Krasnoyarsk, Krasnoyarsk Krai
  - State Budgetary Healthcare Institution "Leningrad Regional Clinical Hospital" ( Site 0588), Gatchina, Leningradskaya Oblast'
  - Russian Scientific Center of Roentgenoradiology ( Site 0559), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 0562), Moscow, Moscow
  - Omsk Clinical Oncology Dispensary ( Site 0568), Omsk, Omsk Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 0576), Samara, Samara Oblast
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0570), Saint Petersburg, Sankt-Peterburg
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 0567), Saint Petersburg, Sankt-Peterburg
  - Tomsk National Scientific Medical Center of Russian Academy of Science ( Site 0579), Tomsk, Tomsk Oblast
- South Korea (5):
  - National Cancer Center ( Site 0174), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0175), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 0176), Songpagu, Seoul
  - Seoul National University Hospital ( Site 0171), Seoul
  - Samsung Medical Center ( Site 0172), Seoul
- Spain (13):
  - Instituto Catalan de Oncologia - ICO ( Site 0330), L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Tauli ( Site 0335), Sabadell, Barcelona
  - Institut Català d'Oncologia (ICO) - Girona ( Site 0321), Girona, Gerona
  - Instituto Valenciano de Oncologia ( Site 0331), Valencia, Valenciana, Comunitat
  - Hospital del Mar ( Site 0333), Barcelona
  - Hospital Provincial San Pedro Alcantara ( Site 0326), Cáceres
  - Hospital Universitario Gregorio Maranon ( Site 0327), Madrid
  - MD Anderson Cancer Center Madrid ( Site 0332), Madrid
  - Hospital Clinico San Carlos ( Site 0324), Madrid
  - Hospital Universitario HM Sanchinarro ( Site 0322), Madrid
  - Hospital Quiron Madrid ( Site 0325), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 0337), Málaga
  - Hospital Virgen del Rocio ( Site 0329), Seville
- Taiwan (5):
  - National Cheng Kung University Hospital ( Site 0134), Tainen, Tainan
  - China Medical University Hospital ( Site 0132), Taichung
  - Taichung Veterans General Hospital ( Site 0133), Taichung
  - National Taiwan University Hospital ( Site 0131), Taipei
  - Taipei Veterans General Hospital ( Site 0135), Taipei
- Turkey (Türkiye) (8):
  - Ege University Medicine of Faculty ( Site 0661), Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCCOLOGY ( Site 0618), Adana
  - Ankara University Hospital Cebeci ( Site 0613), Ankara
  - Hacettepe Universitesi-oncology hospital ( Site 0615), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 0616), Ankara
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Baki-Istanbul Bakirkoy Sadi Konuk Training ( Site 0620), Istanbul
  - Acıbadem Maslak Hastanesi ( Site 0660), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 0619), Istanbul
- Ukraine (8):
  - Cherkasy Regional Oncology Dispensary ( Site 1203), Cherkassy, Cherkasy Oblast
  - Dnepropetrovsk Regional Clinical Hospital Mechnikov-Department of urology ( Site 1205), Dnipro, Dnipropetrovsk Oblast
  - Dnepropetrovsk Regional Clinical Oncology Hospital-Clinical oncological dispensary ( Site 1201), Dnipropetrovsk, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Hospital-Urology department ( Site 1208), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal Non-Commercial Enterprise ""Prykarpatski Clinical Oncological Center"" of Ivano-Frankivsk R ( Site 1209), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNPE Regional Center of Oncology-oncourology department ( Site 1202), Kharkiv, Kharkivs’ka Oblast’
  - LISOD - Israeli Oncological Hospital ""MedX-ray Internationa-Department of Clinical and Scientific ( Site 1207), Kiev, Kyivska Oblast
  - Municipal non-profit enterprise Kyiv City Clinical Oncology -Oncourology department ( Site 1204), Kyiv, Kyivska Oblast
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust ( Site 0530), Bristol, Bristol, City of
  - Cambridge University Hospitals NHS Trust ( Site 0540), Cambridge, Cambridgeshire
  - Torbay Hospital ( Site 0532), Torquay, Devon
  - University College London Hospitals NHS Foundation Trust ( Site 0482), London, London, City of
  - Western General Hospital ( Site 0531), Edinburgh, Midlothian
  - Royal Marsden Hospital (Sutton) ( Site 0526), London, Surrey
  - Musgrove Park Hospital ( Site 0537), Taunton, Worcestershire
  - Mount Vernon Cancer Centre ( Site 0536), Northwood

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Graff JN, Burotto M, Fong PC, Pook DW, Zurawski B, Manneh Kopp R, Salinas J, Bylow KA, Kramer G, Ratta R, Kwiatkowski M, Retz M, Kwak C, Arranz Arija JA, Gurney H, Matsubara N, Villanueva L, Todenhofer T, Liang LW, Todoric J, Imai K, Stenzl A; KEYNOTE-641 Investigators. Pembrolizumab plus enzalutamide versus placebo plus enzalutamide for chemotherapy-naive metastatic castration-resistant prostate cancer: the randomized, double-blind, phase III KEYNOTE-641 study. Ann Oncol. 2025 Aug;36(8):976-987. doi: 10.1016/j.annonc.2025.05.007. Epub 2025 May 16. PMID 40383193
- [Derived] Graff JN, Liang LW, Kim J, Stenzl A. KEYNOTE-641: a Phase III study of pembrolizumab plus enzalutamide for metastatic castration-resistant prostate cancer. Future Oncol. 2021 Aug;17(23):3017-3026. doi: 10.2217/fon-2020-1008. Epub 2021 May 28. PMID 34044584
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://trialstransparency.merckclinicaltrials.com/Study.aspx?id=3475-641&&kw=3475-641

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1244 participants that were randomized to trial, 1235 received treatment. At the time of the primary analysis data cut-off, 635 participants are ongoing in the study.
Groups:
- Pembrolizumab + Enzalutamide: Participants received 200 mg pembrolizumab by intravenous (IV) infusion administered on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 2 years) PLUS enzalutamide 160 mg administered orally (PO) once a day (QD) continuously until progression.
- Placebo + Enzalutamide: Participants received placebo by IV infusion administered on Day 1 Q3W for up to 35 cycles (approximately 2 years) PLUS enzalutamide 160 mg administered PO QD continuously until progression.
Period: Overall Study
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Started | 621 | 623
Treated | 615 | 620
Completed | 0 | 0
Not Completed | 621 | 623
Not completed — Participants Ongoing | 311 | 324
Not completed — Withdrawal by Subject | 20 | 17
Not completed — Physician Decision | 1 | 0
Not completed — Death | 289 | 282

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide | Total
Number analyzed (Participants) | 621 | 623 | 1244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (8.4) | 69.9 (9.1) | 70.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 621 | 623 | 1244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 121 | 126 | 247
  Not Hispanic or Latino | 465 | 466 | 931
  Unknown or Not Reported | 35 | 31 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 12 | 20
  Asian | 80 | 86 | 166
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 12 | 10 | 22
  White | 505 | 494 | 999
  More than one race | 12 | 13 | 25
  Unknown or Not Reported | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS for all participants is presented.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: The efficacy analysis population consisted of all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 24.7 [22.0 to 26.8] | 27.3 [24.5 to 30.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Superiority; p = 0.6621, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.88 to 1.22] — Stratified Cox model with Efron's tie handling method

2. Primary Outcome: Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review
Description: rPFS was defined as the time from randomization to the first documented progressive disease (PD) per PCWG-modified RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurred first. The rPFS per PCWG-modified RECIST for all participants is presented.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 10.4 [8.4 to 12.5] | 9.0 [8.3 to 11.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Superiority; p = 0.4073, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.84 to 1.14] — Stratified Cox model with Efron's tie handling method

3. Secondary Outcome: Time to Initiation of the First Subsequent Anti-cancer Therapy or Death (TFST)
Description: TFST was defined as time from randomization to initiation of the first subsequent anti-cancer therapy or death, whichever occurs first. The TFST for all participants is presented.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 13.2 [11.7 to 15.7] | 12.6 [11.3 to 14.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.83 to 1.09] — Stratified Cox model with Efron's tie handling method

4. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: PSA response rate was defined as percentage of participants in the analysis population who have a negative change (decrease) in PSA level of ≥50% measured twice ≥3 weeks apart. The analysis was performed on participants who had baseline PSA measurements.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: The efficacy analysis population consisted of all randomized participants in the intent to treat population, who had a PSA measurement at baseline, and had data available for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 594 | 601
Percentage of participants | 49.0 [44.9 to 53.1] | 45.1 [41.1 to 49.2]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Difference in Percentage = 3.4, 95% CI 2-sided [-1.5 to 8.3] — Stratified Miettinen and Nurminen method

5. Secondary Outcome: Prostate-specific Antigen (PSA) Undetectable Rate
Description: PSA undetectable rate was defined as percentage of participants in the analysis population with PSA <0.2 ng/mL during study treatment. The analysis was performed on participants who had baseline PSA measurements.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 589 | 596
Percentage of participants | 13.1 [10.5 to 16.1] | 12.6 [10.0 to 15.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Difference in Percentage = 0.3, 95% CI 2-sided [-3.4 to 4.1] — Stratified Miettinen and Nurminen method

6. Secondary Outcome: Objective Response (OR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by as Assessed by Blinded Independent Central Review
Description: OR was defined as the percentage of participants with complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease (NED) on bone scan per PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG).
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Percentage of participants | 12.2 [9.8 to 15.1] | 9.3 [7.1 to 11.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Difference in Percentage = 2.9, 95% CI 2-sided [-0.2 to 6.1] — Stratified Miettinen and Nurminen method

7. Secondary Outcome: Duration of Response (DOR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by as Assessed by Blinded Independent Central Review
Description: DOR was defined as the time from first documented evidence of complete response (CR) or partial response (PR) per PCWG and RECIST 1.1 criteria until progressive disease (PD) or death. PD per RECIST 1.1 was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PD per PCWG was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and were persistent for ≥6 weeks. The DOR was calculated using the product-limit (Kaplan-Meier) method for censored data. If a participant had not progressed, the participant was censored at the date of last disease assessment.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 16.1 [1.4 to 35.3] | 21.5 [0.0 to 35.3]

8. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time from randomization to PSA progression. PSA progression date is defined as the date of 1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, or 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 6.4 [5.5 to 7.1] | 5.6 [4.9 to 6.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.15] — Stratified Cox model with Efron's tie handling method

9. Secondary Outcome: Time to Radiographic Soft Tissue Progression Per Soft Tissue Rules of Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by as Assessed by Blinded Independent Central Review
Description: Time from randomization to radiographic soft tissue progression per PCWG-modified RECIST 1.1
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | 20.7 [18.0 to 30.1] | 26.3 [17.8 to NA] — NA= Upper limit not reached at time of data cut off
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.74 to 1.09] — Stratified Cox model with Efron's tie handling method

10. Secondary Outcome: Time to Pain Progression (TTPP) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("Worst Pain in 24 Hours") and Opiate Analgesic Use (Analgesic Quantification Algorithm [AQA] Score)
Description: Time from randomization to pain progression. In this study, pain progression was assessed by participant responses to Item 3 of the BPI-SF and participant AQA Scores which are both assessed by participants daily for 7 consecutive days.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: All participants in the patient-reported outcomes (PRO) full analysis set who received at least 1 dose of study treatment and who had at least 1 PRO assessment available. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 612 | 618
Months | NA [23.3 to NA] — NA= Median and upper limit not reached at time of data cut off | NA [NA to NA] — NA= Median, lower limit, and upper limit not reached at time of data cut off
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.82 to 1.35] — Stratified Cox model with Efron's tie handling method

11. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (SSRE)
Description: Time from randomization to the first SSRE. SSRE is defined as radiation to prevent or relieve skeletal symptoms, occurrence of new symptomatic pathological fracture, spinal cord compression, or surgery to bone.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 621 | 623
Months | NA [NA to NA] — NA= Median, lower limit, and upper limit not reached at time of data cut off | NA [NA to NA] — NA= Median, lower limit, and upper limit not reached at time of data cut off
Statistical Analysis 1: Comparison: Pembrolizumab + Enzalutamide vs Placebo + Enzalutamide; Test type: Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.85 to 1.51] — Stratified Cox model with Efron's tie handling method

12. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants who experienced an AE is presented.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 615 | 620
Participants | 594 | 596

13. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide
Number analyzed (Participants) | 615 | 620
Participants | 115 | 50

ADVERSE EVENTS:
Time Frame: Up to 40 months (through database cut-off date of 12-Dec-2022)
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) include all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", and "Disease progression" not related to study drug are excluded as AEs. Data are reported by treatment received.
Groups:
- Pembrolizumab + Enzalutamide Second Course: Qualified participants who received pembrolizumab as a first course and stopped the first course of pembrolizumab due to complete response (CR) or completed the first course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional) plus enzalutamide.
Arm/Group | Pembrolizumab + Enzalutamide | Placebo + Enzalutamide | Pembrolizumab + Enzalutamide Second Course
All-Cause Mortality (participants affected / at risk) | 295/621 | 291/623 | 1/4
Serious Adverse Events (participants affected / at risk) | 238/615 | 165/620 | 0/4
Other Adverse Events (participants affected / at risk) | 563/615 | 551/620 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide (N=615) | Placebo + Enzalutamide (N=620) | Pembrolizumab + Enzalutamide Second Course (N=4)
Acquired factor VIII deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 4 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 6 (6) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Primary adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 3 (3) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 7 (7) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cytomegalovirus gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 16 (16) | 10 (12) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 10 (13) | 0 (0)
Urosepsis (Infections and infestations) | 8 (8) | 3 (3) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postpolypectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
T-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mononeuropathy multiplex (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 9 (9) | 11 (11) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 10 (11) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 5 (5) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Enzalutamide (N=615) | Placebo + Enzalutamide (N=620) | Pembrolizumab + Enzalutamide Second Course (N=4)
Anaemia (Blood and lymphatic system disorders) | 141 (201) | 103 (119) | 0 (0)
Hypothyroidism (Endocrine disorders) | 76 (81) | 27 (28) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 25 (27) | 34 (41) | 0 (0)
Constipation (Gastrointestinal disorders) | 113 (124) | 90 (109) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 115 (153) | 79 (104) | 0 (0)
Nausea (Gastrointestinal disorders) | 126 (150) | 114 (139) | 0 (0)
Vomiting (Gastrointestinal disorders) | 54 (64) | 34 (45) | 0 (0)
Asthenia (General disorders) | 109 (124) | 97 (111) | 0 (0)
Fatigue (General disorders) | 190 (213) | 170 (186) | 0 (0)
Oedema peripheral (General disorders) | 46 (54) | 42 (43) | 0 (0)
Pyrexia (General disorders) | 46 (56) | 22 (24) | 0 (0)
COVID-19 (Infections and infestations) | 52 (54) | 35 (35) | 0 (0)
Urinary tract infection (Infections and infestations) | 40 (52) | 44 (57) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 33 (44) | 28 (33) | 0 (0)
Alanine aminotransferase increased (Investigations) | 34 (38) | 24 (27) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 40 (49) | 32 (39) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 33 (41) | 24 (25) | 0 (0)
Blood creatinine increased (Investigations) | 31 (38) | 24 (32) | 0 (0)
Weight decreased (Investigations) | 90 (92) | 73 (74) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 146 (167) | 124 (136) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 31 (44) | 24 (31) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 149 (201) | 128 (167) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 120 (142) | 123 (140) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 39 (42) | 52 (57) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 26 (29) | 32 (35) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 34 (35) | 30 (33) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 54 (59) | 60 (73) | 0 (0)
Dizziness (Nervous system disorders) | 44 (47) | 44 (49) | 0 (0)
Headache (Nervous system disorders) | 49 (63) | 55 (66) | 0 (0)
Insomnia (Psychiatric disorders) | 30 (32) | 52 (54) | 0 (0)
Haematuria (Renal and urinary disorders) | 43 (50) | 42 (47) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (41) | 21 (22) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 32 (37) | 23 (24) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 95 (115) | 44 (47) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 139 (184) | 43 (51) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 42 (50) | 8 (9) | 0 (0)
Hot flush (Vascular disorders) | 39 (42) | 49 (51) | 0 (0)
Hypertension (Vascular disorders) | 64 (77) | 72 (89) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03834493/Prot_SAP_000.pdf